CLINICAL TRIAL: NCT04176939
Title: Long-term Immunogenicity Study of Herpes Zoster Subunit Vaccine (GSK1437173A) and Immunogenicity and Safety Assessment of Revaccination With Two Additional Doses in Adults With Renal Transplant From Study ZOSTER-041
Brief Title: A Study to Test GlaxoSmithKline's (GSK) Herpes Zoster (HZ) Subunit Vaccine's Long-term Immune Response in Previously Vaccinated Kidney Transplant Adults and Then to Test if 2 Additional Doses of the Vaccine Are Safe and Able to Generate an Immune Response
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 212340; 2019-001815-21 (EudraCT Number)
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HZ/su Group (Experimental): Participants with renal transplant who completed the 2-dose Herpes Zoster (HZ/su) vaccination course in the primary ZOSTER-041 (NCT02058589) study were enrolled in the current ZOSTER-073 (NCT04176939) study.
  47 of these participants further received 1 or 2 additional doses of HZ/su vaccine in the revaccination phase of the current ZOSTER-073 (NCT04176939) study, first dose at Month 24 and second dose at Month 25.
  Interventions: Biological: HZ/su vaccine (GSK1437173A)

INTERVENTIONS:
Biological: HZ/su vaccine (GSK1437173A) — 2 intramuscular (IM) revaccination doses of the HZ/su vaccine administered - first dose at Month 24 and second dose at Month 25.

SUMMARY:
The purpose of this study was to evaluate the long-term immune responses to the Herpes Zoster subunit (HZ/su) vaccine as well as safety up to 7 years after the 2-dose primary vaccination course from study ZOSTER-041 (NCT02058589). This study also assessed immune responses as well as safety after revaccination with 2 additional doses of the HZ/su administered at 6 to 8 years after the 2-dose primary vaccination course.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for enrolment

  * Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol or/and subjects' Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
  * Written informed consent obtained from the subject/LAR(s) of the subject prior to performance of any study-specific procedure.
  * Subjects who previously participated in study ZOSTER-041 and completed the full 2 dose HZ/su primary vaccination course.
* Inclusion criteria for revaccination

  * Subjects receiving maintenance CIS therapy for the prevention of allograft rejection for a minimum of one month prior to the first revaccination.
  * Subjects without an episode of allograft rejection within 90 days prior to the first revaccination visit.
  * Female subjects of non-childbearing potential may be revaccinated. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
  * Female subjects of childbearing potential may be revaccinated, if the subject:
* has practiced adequate contraception for 30 days prior to revaccination, and
* has a negative pregnancy test on the day of revaccination, and
* has agreed to continue adequate contraception up to 2 months after completion of the revaccination series.

Exclusion Criteria:

Exclusion criteria for enrolment Medical conditions

* Vaccination against HZ since completion of study ZOSTER-041.
* Significant underlying illness that, in the opinion of the investigator, is expected to prevent completion of the study.
* Any other condition that, in the opinion of the investigator, would interfere with the evaluations required by the study.

Prior/Concurrent clinical study experience

• Concurrently participating in another interventional vaccine or immunosuppressive clinical study, in which the subject is exposed to an investigational or a non-investigational vaccine/product (drug) at any time during the ZOSTER-073 study.

Exclusion criteria for revaccination Medical conditions

* History of confirmed HZ within one year before revaccination visit (Visit 3).
* More than one organ transplanted.
* Any additional confirmed or suspected immunosuppressive or immunodeficient condition.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Any other condition that, in the opinion of the investigator, would interfere with the evaluations required by the study or make vaccination unsafe.

Prior/Concomitant therapy

* Administration or planned administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the first revaccination dose of study vaccine and ending at Visit 5 (Month 26).
* Use of anti-CD20 or other B-cell monoclonal antibody agents as maintenance and/or therapeutic immunosuppressive therapy for the prevention of allograft rejection within 9 months of first revaccination dose of study vaccine.
* Evidence or high suspicion, in the opinion of the investigator, of noncompliance or nonadherence to use of maintenance immunosuppressive therapies.
* Planned administration/administration of a live vaccine in the period starting 30 days before the first dose and ending 30 days after the last dose of study vaccine administration.
* Planned administration/administration of a non-replicating or subunit vaccine, not foreseen by the study protocol, in the period starting 8 days before and ending 30 days after each dose of study vaccine.

Other exclusion criteria for revaccination

* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions up to 2 months post-revaccination Dose 2.
* Any condition which, in the judgment of the investigator, would make intramuscular injection unsafe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- GSK Investigational Site, Brussels, Belgium
- GSK Investigational Site, Toronto, Ontario, Canada
- GSK Investigational Site, Helsinki, Finland
- GSK Investigational Site, Panama City, Panama
- GSK Investigational Site, Seoul, South Korea
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
- GSK Investigational Site, Tau-Yuan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants from the Herpes Zoster (HZ/su) treatment group of ZOSTER-041 (NCT02058589) study who had a complete primary vaccination course (2 doses of HZ/su vaccine) were offered enrollment in the current ZOSTER-073 study (NCT04176939). A total of 68 participants met the eligibility criteria and consented to participate in this study.
Pre-assignment Details: Out of the 68 participants originally enrolled in the current ZOSTER-073 study (Enrolled Set), 21 participants did not receive any revaccination doses, hence only 47 participants were vaccinated with at least one revaccination dose and included in the Exposed Set for revaccination phase in this study.
Period: Overall Study
Arm/Group | HZ/su Group
Started (Started = number of participants enrolled in the study (Enrolled Set)) | 68
Revaccinated (Revaccinated = number of participants included in the Exposed Set for revaccination phase) | 47
Completed | 49
Not Completed | 19
Not completed — Withdrawal by Subject | 5
Not completed — Migrated / Moved From The Study Area | 1
Not completed — Lost to Follow-up | 2
Not completed — Unspecified reason | 4
Not completed — Adverse Event Requiring Expedited Reporting | 7

BASELINE CHARACTERISTICS:
Arm/Group | HZ/su Group
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] — Descriptive summaries of Age at the time of enrollment in the current ZOSTER-073 study are presented for the participants enrolled in this study (Enrolled Set).
  Years | 58.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Descriptive summaries of Sex at the time of enrollment in the current ZOSTER-073 study are presented for the participants enrolled in this study (Enrolled Set).
  Participants
    Female | 22
    Male | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Descriptive summaries of Race/Ethnicity at the time of enrollment in the current ZOSTER-073 study are presented for the participants enrolled in this study (Enrolled Set).
  Participants
    ASIAN | 14
    BLACK OR AFRICAN AMERICAN | 3
    WHITE | 46
    OTHER - UNSPECIFIED | 5

OUTCOME MEASURES:

1. Primary Outcome: Anti-glycoprotein E (Anti-gE) Antibody Concentrations, as Assessed in the Long Term Follow-up (LTFU) Phase of the Current ZOSTER-073 Study
Description: Anti-gE antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs) in milli-international units per milliliter (mIU/mL).
Time Frame: At Day 1, Month 12 and Month 24 (pre-revaccination) in the current ZOSTER-073 study
Population: Analysis was performed on the Per Protocol Set for analysis of persistence (LTFU phase), which included evaluable participants from the Enrolled Set with a complete vaccination course (2 doses of HZ/su vaccine) in the ZOSTER-041 study, who met the eligibility criteria and signed informed consent in the current study and for whom persistence immunogenicity results after primary vaccination course were available at the specified time points in the current study, regardless of revaccination status.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HZ/su Group
Number analyzed (Participants) | 60
mIU/mL
  At Day 1: number analyzed (Participants) | 56
  At Day 1 | 3729.8 [2736.2 to 5084.0]
  At Month 12 | 3440.2 [2499.0 to 4735.7]
  At Month 24: number analyzed (Participants) | 49
  At Month 24 | 3075.8 [2091.8 to 4522.8]

2. Primary Outcome: Anti-gE Antibody Concentrations, as Assessed in the Revaccination Active Phase of the Current ZOSTER-073 Study
Description: Anti-gE antibody concentrations were determined by ELISA and expressed as GMCs in mIU/mL.
Time Frame: At Month 24 (pre-revaccination), Month 25 (1 month post-revaccination Dose 1) and Month 26 (1 month post-revaccination Dose 2) in the current ZOSTER-073 study
Population: Analysis was performed on the Per Protocol Set for Immunogenicity after revaccination course (Revaccination active phase), which included evaluable participants who were administered 1 or 2 doses of revaccination as per the revaccination schedule and who had immunogenicity data available for the specified analysis at the specified time points in the current study.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HZ/su Group
Number analyzed (Participants) | 45
mIU/mL
  At Month 24 | 2828.5 [1886.6 to 4240.5]
  At Month 25: number analyzed (Participants) | 44
  At Month 25 | 27655.5 [17882.7 to 42769.1]
  At Month 26: number analyzed (Participants) | 44
  At Month 26 | 31517.0 [21581.1 to 46027.3]

3. Secondary Outcome: Frequency of gE-specific Cluster of Differentiation 4 (CD4) (2+) T-cells, as Assessed in the LTFU Phase of the Current ZOSTER-073 Study
Description: Frequency of gE-specific CD4 (2+) T-cells expressing two or more activation markers (from among interferon gamma [IFN-γ], interleukin-2 [IL-2], tumour necrosis factor alpha [TNF-α] and CD40 Ligand [CD40L]) was determined by intracellular cytokine staining (ICS) as measured by cytokine flow cytometry (CFC) and expressed in CD4(2+) T-cells per million cells [CD4(2+) T-cells/million cells].
Time Frame: At Day 1, Month 12 and Month 24 (pre-revaccination) in the current ZOSTER-073 study
Population: Analysis was performed on a sub-cohort of participants from the Per Protocol Set for analysis of persistence (LTFU phase), for whom an additional blood sample for cell-mediated immunity (CMI) analysis was collected and who had CMI results available for the specified analysis at the specified time points in the current study.
Measure: Median (Inter-Quartile Range); unit: CD4(2+) T-cells/million cells
Arm/Group | HZ/su Group
Number analyzed (Participants) | 28
CD4(2+) T-cells/million cells
  At Day 1 | 608.9 [167.2 to 993.6]
  At Month 12: number analyzed (Participants) | 18
  At Month 12 | 299.4 [105.3 to 1068.4]
  At Month 24: number analyzed (Participants) | 19
  At Month 24 | 711.0 [309.9 to 1211.0]

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) Related to Primary Vaccination in ZOSTER-041 Study, as Assessed in the LTFU Phase of the Current ZOSTER-073 Study
Description: SAEs assessed included any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization or resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study participant. SAEs related to primary vaccination in ZOSTER-041 study were assessed by the investigator.
Time Frame: From Month 13 (last visit) in ZOSTER-041 study until Month 24 in the current ZOSTER-073 study
Population: Analysis was performed on the Enrolled Set, which included all participants with a complete vaccination course (2 doses of HZ/su vaccine) in ZOSTER-041 study who met the eligibility criteria and signed informed consent in the current study.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 68
Participants | 0

5. Secondary Outcome: Number of Participants With Suspected or Confirmed Herpes Zoster (HZ) Cases, as Assessed in the LTFU Phase of the Current ZOSTER-073 Study
Description: A suspected HZ case was defined as a new unilateral rash accompanied by pain (broadly defined to include allodynia, pruritus or other sensations) without alternative diagnosis.
  A confirmed HZ case was diagnosed by an algorithm that included Polymerase Chain Reaction (PCR) and the HZ Ascertainment Committee (HZAC) determination.
Time Frame: From Month 13 (last visit) in ZOSTER-041 study until Day 1 (first visit) in the current ZOSTER-073 study
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 68
Participants
  Confirmed HZ case | 0
  Suspected HZ case | 3

6. Secondary Outcome: Number of Participants With Confirmed HZ Cases, as Assessed in the LTFU Phase of the Current ZOSTER-073 Study
Description: A confirmed HZ case was diagnosed by an algorithm that included Polymerase Chain Reaction (PCR) and the HZ Ascertainment Committee (HZAC) determination.
Time Frame: From Day 1 until Month 24 in the current ZOSTER-073 study
Population: Analysis was performed on the Enrolled Set, which included all participants with a complete vaccination course (2 doses of HZ/su vaccine) in ZOSTER-041 primary study who met the eligibility criteria and signed informed consent in the current study.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 68
Participants | 3

7. Secondary Outcome: Number of Participants With Suspected or Biopsy-proven Allograft Rejections, as Assessed in the LTFU Phase of the Current ZOSTER-073 Study
Description: The number of participants with biopsy for clinical indication (suspected) or surveillance protocol that was not biopsy-proven rejection and with biopsy-proven allograft rejections are reported. Biopsy-proven allograft rejections are defined as adverse events of specific interest (AESIs).
Time Frame: From Month 13 (last visit) in ZOSTER-041 study until Day 1 (first visit) in the current ZOSTER-073 study
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 68
Participants
  Biopsy-proven allograft rejection | 0
  Biopsy for clinical indication (suspected) or surveillance protocol | 5

8. Secondary Outcome: Number of Participants With Biopsy-proven Allograft Rejections, as Assessed in the LTFU Phase of the Current ZOSTER-073 Study
Description: Biopsy-proven allograft rejection is defined as an adverse event of specific interest (AESI).
Time Frame: From Day 1 until Month 24 in the current ZOSTER-073 study
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 68
Participants | 2

9. Secondary Outcome: Number of Participants With Allograft Dysfunction Related to Allograft Rejection Episodes, as Assessed in the LTFU Phase of the Current ZOSTER-073 Study
Description: Declining allograft function (allograft dysfunction) was assessed through all clinically obtained serum creatinine values from 2 months prior to an episode of biopsy-proven rejection and up to 2 months after rejection resolution and cessation of therapeutic immunosuppressive therapy. Allograft dysfunction is defined as having a fold increase in serum creatinine of 1.2 greater from the reference timepoint (2 months prior to an episode of biopsy-proven rejection).
Time Frame: From Month 13 (last visit) in ZOSTER-041 study until Month 24 in the current ZOSTER-073 study
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 68
Participants | 0

10. Secondary Outcome: Number of Participants With Allograft Dysfunction Related to HZ Episodes, as Assessed in the LTFU Phase of the Current ZOSTER-073 Study
Description: Declining allograft function was assessed through all clinically obtained serum creatinine values from 2 months prior to an episode of HZ and up to 2 months after HZ rash resolution. Allograft dysfunction is defined as having a fold increase in serum creatinine of 1.2 greater from the reference timepoint (2 months prior to an episode of HZ).
Time Frame: From Month 13 (last visit) in ZOSTER-041 study until Month 24 in the current ZOSTER-073 study
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 68
Participants | 0

11. Secondary Outcome: Frequency of gE-specific CD4(2+) T-cells, as Assessed in the Revaccination Active Phase of the Current ZOSTER-073 Study
Description: Frequency of gE-specific CD4 (2+) T-cells expressing two or more activation markers (from among IFN-γ, IL-2, TNF-α and CD40L) was determined by ICS as measured by CFC and expressed in CD4(2+) T-cells/million cells.
Time Frame: as for outcome 2
Population: Analysis was performed on a sub-cohort of participants from the Per Protocol Set for Immunogenicity after revaccination course (Revaccination active phase), for whom an additional blood sample for CMI analysis was collected and who had CMI results available for the specified analysis at the specified time points in the current study.
Measure: Median (Inter-Quartile Range); unit: CD4(2+) T-cells/million cells
Arm/Group | HZ/su Group
Number analyzed (Participants) | 23
CD4(2+) T-cells/million cells
  At Month 24 | 793.5 [309.9 to 1235.8]
  At Month 25: number analyzed (Participants) | 20
  At Month 25 | 4476.2 [3136.7 to 7704.6]
  At Month 26: number analyzed (Participants) | 18
  At Month 26 | 3747.3 [2758.1 to 8906.2]

12. Secondary Outcome: Anti-gE Antibody Concentrations, as Assessed in the Revaccination Follow-up Phase of the Current ZOSTER-073 Study
Description: Persistence of humoral immunity after the revaccination course was evaluated in terms of anti-gE antibody concentrations. Anti-gE antibody concentrations were determined by ELISA and expressed as GMCs in mIU/mL.
Time Frame: At Month 37 (12 months post-revaccination Dose 2) and Month 49 (24 months post-revaccination Dose 2) in the current ZOSTER-073 study
Population: Analysis was performed on the Per Protocol Set for persistence after revaccination course (Revaccination follow-up phase), which included evaluable participants who received 2 doses of revaccination in the current ZOSTER-073 study and for whom immunogenicity persistence results after revaccination were available for the specified analysis at the specified time points in the current study.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HZ/su Group
Number analyzed (Participants) | 44
mIU/mL
  At Month 37 | 23989.4 [17539.6 to 32811.0]
  At Month 49: number analyzed (Participants) | 36
  At Month 49 | 9985.8 [5917.8 to 16850.0]

13. Secondary Outcome: Frequency of gE-specific CD4(2+) T-cells, as Assessed in the Revaccination Follow-up Phase of the Current ZOSTER-073 Study
Description: as for outcome 11
Time Frame: as for outcome 12
Population: Analysis was performed on a sub-cohort of participants from the Per Protocol Set for persistence after revaccination course (Revaccination follow-up phase), for whom an additional blood sample for CMI analysis was collected and who had CMI results available for the specified analysis at the specified time points in the current study.
Measure: Median (Inter-Quartile Range); unit: CD4(2+) T-cells/million cells
Arm/Group | HZ/su Group
Number analyzed (Participants) | 20
CD4(2+) T-cells/million cells
  At Month 37 | 1777.4 [1297.7 to 2505.4]
  At Month 49: number analyzed (Participants) | 16
  At Month 49 | 1144.9 [818.1 to 2724.1]

14. Secondary Outcome: Number of Participants With Any and Grade 3 Solicited Administration Site Events After Each Revaccination, as Assessed in the Revaccination Active Phase of the Current ZOSTER-073 Study
Description: Assessed solicited administration site events included erythema, pain and swelling at injection site. Any = occurrence of the event regardless of intensity grade. Any erythema/swelling at injection site = erythema/swelling at injection site with a diameter larger than (>) 20 millimeters (mm). Grade 3 pain = significant pain at rest, which prevented normal, everyday activities. Grade 3 erythema/swelling at injection site = erythema/swelling at injection site with a diameter >100 mm.
Time Frame: Within 7 days after each revaccination dose (administered at Month 24 [Dose 1] and at Month 25 [Dose 2]) in the current ZOSTER-073 study
Population: Analysis was performed on the Exposed Set for revaccination phase, which included all participants with at least one HZ/su revaccination dose administered in the current study and with the solicited administration site events diary card data available after the corresponding revaccination, for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 45
Participants
  Any Erythema, after revaccination Dose 1 | 9
  Grade 3 Erythema, after revaccination Dose 1 | 0
  Any Erythema, after revaccination Dose 2 | 6
  Grade 3 Erythema, after revaccination Dose 2 | 0
  Any Pain, after revaccination Dose 1 | 37
  Grade 3 Pain, after revaccination Dose 1 | 7
  Any Pain, after revaccination Dose 2 | 31
  Grade 3 Pain, after revaccination Dose 2 | 2
  Any Swelling, after revaccination Dose 1 | 7
  Grade 3 Swelling, after revaccination Dose 1 | 0
  Any Swelling, after revaccination Dose 2 | 4
  Grade 3 Swelling, after revaccination Dose 2 | 0

15. Secondary Outcome: Duration in Days of Solicited Administration Site Events After Each Revaccination, as Assessed in the Revaccination Active Phase of the Current ZOSTER-073 Study
Description: Duration is the number of days in which a participant experienced the solicited administration site event within the 7-day solicited follow-up period. Assessed solicited administration site events included erythema, pain and swelling at injection site.
Time Frame: as for outcome 14
Population: Analysis was performed on the Exposed Set for revaccination phase, which included participants with at least one HZ/su revaccination dose administered in the current study, with solicited diary data available after the corresponding revaccination, who experienced the specified solicited administration site event within 7 days following the respective revaccination dose and with the duration documented.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | HZ/su Group
Number analyzed (Participants) | 37
Days
  Erythema, after revaccination Dose 1: number analyzed (Participants) | 9
  Erythema, after revaccination Dose 1 | 4.0 [1.0 to 5.0]
  Pain, after revaccination Dose 1 | 3.0 [2.0 to 4.0]
  Swelling, after revaccination Dose 1: number analyzed (Participants) | 6
  Swelling, after revaccination Dose 1 | 3.0 [2.0 to 3.0]
  Erythema, after revaccination Dose 2: number analyzed (Participants) | 6
  Erythema, after revaccination Dose 2 | 3.0 [2.0 to 3.0]
  Pain, after revaccination Dose 2: number analyzed (Participants) | 31
  Pain, after revaccination Dose 2 | 2.0 [2.0 to 3.0]
  Swelling, after revaccination Dose 2: number analyzed (Participants) | 4
  Swelling, after revaccination Dose 2 | 2.5 [1.5 to 3.5]

16. Secondary Outcome: Number of Participants With Any, Grade 3 and Related Solicited Systemic Events After Each Revaccination, as Assessed in the Revaccination Active Phase of the Current ZOSTER-073 Study
Description: Assessed solicited systemic events included fatigue, gastrointestinal symptoms (including nausea, vomiting, diarrhea and/or abdominal pain), headache, myalgia, shivering and fever [temperature higher than or equal (>=) to 38.0 degrees Celsius (°C)/100.4 degrees Fahrenheit (°F)]. Any AE = occurrence of the event regardless of intensity grade. Grade 3 fatigue, gastrointestinal symptoms, headache, myalgia, shivering = event that prevented normal, everyday activities. Grade 3 fever = temperature higher (>) than 39°C/102.2°F. Related fatigue, gastrointestinal symptoms, headache, myalgia, shivering, fever = event assessed by the investigator as related to the revaccination. The preferred route for measuring temperature in this study was oral.
Time Frame: as for outcome 14
Population: Analysis was performed on the Exposed Set for revaccination phase, which included all participants with at least one HZ/su revaccination dose administered in the current study and with the solicited systemic events diary card data available after the corresponding revaccination, for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 46
Participants
  Any Fatigue, after revaccination Dose 1 | 26
  Grade 3 Fatigue, after revaccination Dose 1 | 2
  Related Fatigue, after revaccination Dose 1 | 22
  Any Fatigue, after revaccination Dose 2: number analyzed (Participants) | 45
  Any Fatigue, after revaccination Dose 2 | 23
  Grade 3 Fatigue, after revaccination Dose 2: number analyzed (Participants) | 45
  Grade 3 Fatigue, after revaccination Dose 2 | 2
  Related Fatigue, after revaccination Dose 2: number analyzed (Participants) | 45
  Related Fatigue, after revaccination Dose 2 | 21
  Any Gastrointestinal symptoms, after revaccination Dose 1 | 11
  Grade 3 Gastrointestinal symptoms, after revaccination Dose 1 | 0
  Related Gastrointestinal symptoms, after revaccination Dose 1 | 10
  Any Gastrointestinal symptoms, after revaccination Dose 2: number analyzed (Participants) | 45
  Any Gastrointestinal symptoms, after revaccination Dose 2 | 10
  Grade 3 Gastrointestinal symptoms, after revaccination Dose 2: number analyzed (Participants) | 45
  Grade 3 Gastrointestinal symptoms, after revaccination Dose 2 | 1
  Related Gastrointestinal symptoms, after revaccination Dose 2: number analyzed (Participants) | 45
  Related Gastrointestinal symptoms, after revaccination Dose 2 | 9
  Any Headache, after revaccination Dose 1 | 22
  Grade 3 Headache, after revaccination Dose 1 | 3
  Related Headache, after revaccination Dose 1 | 19
  Any Headache, after revaccination Dose 2: number analyzed (Participants) | 45
  Any Headache, after revaccination Dose 2 | 16
  Grade 3 Headache, after revaccination Dose 2: number analyzed (Participants) | 45
  Grade 3 Headache, after revaccination Dose 2 | 0
  Related Headache, after revaccination Dose 2: number analyzed (Participants) | 45
  Related Headache, after revaccination Dose 2 | 16
  Any Myalgia, after revaccination Dose 1 | 21
  Grade 3 Myalgia, after revaccination Dose 1 | 1
  Related Myalgia, after revaccination Dose 1 | 17
  Any Myalgia, after revaccination Dose 2: number analyzed (Participants) | 45
  Any Myalgia, after revaccination Dose 2 | 19
  Grade 3 Myalgia, after revaccination Dose 2: number analyzed (Participants) | 45
  Grade 3 Myalgia, after revaccination Dose 2 | 1
  Related Myalgia, after revaccination Dose 2: number analyzed (Participants) | 45
  Related Myalgia, after revaccination Dose 2 | 16
  Any Shivering, after revaccination Dose 1 | 15
  Grade 3 Shivering, after revaccination Dose 1 | 3
  Related Shivering, after revaccination Dose 1 | 13
  Any Shivering, after revaccination Dose 2: number analyzed (Participants) | 45
  Any Shivering, after revaccination Dose 2 | 10
  Grade 3 Shivering, after revaccination Dose 2: number analyzed (Participants) | 45
  Grade 3 Shivering, after revaccination Dose 2 | 1
  Related Shivering, after revaccination Dose 2: number analyzed (Participants) | 45
  Related Shivering, after revaccination Dose 2 | 9
  Any Fever, after revaccination Dose 1 | 4
  Grade 3 Fever, after revaccination Dose 1 | 1
  Related Fever, after revaccination Dose 1 | 4
  Any Fever, after revaccination Dose 2: number analyzed (Participants) | 45
  Any Fever, after revaccination Dose 2 | 4
  Grade 3 Fever, after revaccination Dose 2: number analyzed (Participants) | 45
  Grade 3 Fever, after revaccination Dose 2 | 1
  Related Fever, after revaccination Dose 2: number analyzed (Participants) | 45
  Related Fever, after revaccination Dose 2 | 4

17. Secondary Outcome: Duration in Days of Solicited Systemic Events After Each Revaccination, as Assessed in the Revaccination Active Phase of the Current ZOSTER-073 Study
Description: Duration is the number of days in which a participant experienced the solicited systemic event within the 7-day solicited follow-up period. Assessed solicited systemic events included fatigue, gastrointestinal symptoms (including nausea, vomiting, diarrhea and/or abdominal pain), headache, myalgia, shivering and fever.
Time Frame: as for outcome 14
Population: Analysis was performed on the Exposed Set for revaccination phase, which included participants with at least one HZ/su revaccination dose administered in the current study, with solicited diary data available after the corresponding revaccination, who experienced the specified solicited systemic event within 7 days following the respective revaccination dose and with the duration documented.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | HZ/su Group
Number analyzed (Participants) | 26
Days
  Fatigue, after revaccination Dose 1 | 3.0 [2.0 to 3.0]
  Gastrointestinal symptoms, after revaccination Dose 1: number analyzed (Participants) | 11
  Gastrointestinal symptoms, after revaccination Dose 1 | 2.0 [1.0 to 2.0]
  Headache, after revaccination Dose 1: number analyzed (Participants) | 22
  Headache, after revaccination Dose 1 | 2.0 [1.0 to 3.0]
  Myalgia, after revaccination Dose 1: number analyzed (Participants) | 21
  Myalgia, after revaccination Dose 1 | 2.0 [2.0 to 4.0]
  Shivering, after revaccination Dose 1: number analyzed (Participants) | 15
  Shivering, after revaccination Dose 1 | 1.0 [1.0 to 2.0]
  Fever, after revaccination Dose 1: number analyzed (Participants) | 4
  Fever, after revaccination Dose 1 | 1.5 [1.0 to 2.0]
  Fatigue, after revaccination Dose 2: number analyzed (Participants) | 23
  Fatigue, after revaccination Dose 2 | 2.0 [2.0 to 4.0]
  Gastrointestinal symptoms, after revaccination Dose 2: number analyzed (Participants) | 10
  Gastrointestinal symptoms, after revaccination Dose 2 | 1.5 [1.0 to 2.0]
  Headache, after revaccination Dose 2: number analyzed (Participants) | 16
  Headache, after revaccination Dose 2 | 2.0 [1.0 to 3.0]
  Myalgia, after revaccination Dose 2: number analyzed (Participants) | 19
  Myalgia, after revaccination Dose 2 | 2.0 [1.0 to 4.0]
  Shivering, after revaccination Dose 2: number analyzed (Participants) | 10
  Shivering, after revaccination Dose 2 | 2.0 [1.0 to 2.0]
  Fever, after revaccination Dose 2: number analyzed (Participants) | 4
  Fever, after revaccination Dose 2 | 1.0 [1.0 to 1.0]

18. Secondary Outcome: Number of Participants With Any, Grade 3 and Related Unsolicited Adverse Events (AEs) Post-revaccination, as Assessed in the Revaccination Active Phase of the Current ZOSTER-073 Study
Description: An unsolicited AE was defined as any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited AE. Any = occurrence of the event regardless of intensity grade or relation to revaccination. Grade 3 = event that prevented normal, everyday activities. Related = event assessed by the investigator as related to revaccination.
Time Frame: Within 30 days (across revaccination doses) post-revaccination period in the current ZOSTER-073 study
Population: Analysis was performed on the Exposed Set for revaccination phase, which included all participants with at least one HZ/su revaccination dose administered in the current study and for whom unsolicited AEs data were available for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 47
Participants
  Any unsolicited AE(s) | 12
  Grade 3 unsolicited AE(s) | 3
  Related unsolicited AE(s) | 2

19. Secondary Outcome: Number of Participants With Any Serious Adverse Events (SAEs) and Fatal SAEs, as Assessed in the Revaccination Active Phase of the Current ZOSTER-073 Study
Description: SAEs assessed included any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization or resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study participant. Any = occurrence of the SAE regardless of intensity grade or relation to revaccination. Fatal = SAE resulting in the death of the participant.
Time Frame: From Month 24 (pre-revaccination) until Month 37 (12 months post-revaccination Dose 2) in the current ZOSTER-073 study
Population: Analysis was performed on the Exposed Set for revaccination phase, which included all participants with at least one HZ/su revaccination dose administered in the current study and for whom SAEs data were available for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 47
Participants
  Any SAE(s) | 9
  Fatal SAE(s) | 1

20. Secondary Outcome: Number of Participants With Related SAEs and Related-fatal SAEs, as Assessed in the Revaccination Active Phase of the Current ZOSTER-073 Study
Description: SAEs assessed included any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization or resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study participant. Related = SAE assessed by the investigator as related to revaccination. Related-fatal = SAE resulting in the death of the participant assessed by the investigator as related to revaccination.
Time Frame: From Month 24 (pre-revaccination) until Month 49 (24 months post-revaccination Dose 2) in the current ZOSTER-073 study
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 47
Participants
  Related SAE(s) | 0
  Related-fatal SAE(s) | 0

21. Secondary Outcome: Number of Participants With Any and Related Biopsy-proven Allograft Rejections, as Assessed in the Revaccination Active and Follow-up Phases of the Current ZOSTER-073 Study
Description: Biopsy-proven allograft rejection is defined as an adverse event of special interest (AESI) and is recorded in serious adverse event (SAE) screens, irrespective of the seriousness of the event. Related biopsy proven allograft rejections = biopsy-proven allograft rejections assessed by the investigator as related to revaccination.
Time Frame: From Month 24 (pre-revaccination) until Month 49 (24 months post-revaccination Dose 2) in the current ZOSTER-073 study
Population: Analysis was performed on the Exposed Set for revaccination phase, which included all participants with at least one HZ/su revaccination dose administered in the current study and for whom biopsy-proven allograft rejections data were available for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 47
Participants
  Any biopsy-proven allograft rejection | 1
  Related biopsy-proven allograft rejection | 0

22. Secondary Outcome: Number of Participants With Any and Related Potential Immune-mediated Diseases (pIMDs), as Assessed in the Revaccination Active and Follow-up Phases of the Current ZOSTER-073 Study
Description: pIMDs are defined as a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology. Any = occurrence of the pIMD regardless of intensity grade or relation to revaccination. Related = pIMDs assessed by the investigator as related to revaccination.
Time Frame: From Month 24 (pre-revaccination) until Month 37 (12 months post-revaccination Dose 2) in the current ZOSTER-073 study
Population: Analysis was performed on the Exposed Set for revaccination phase, which included all participants with at least one HZ/su revaccination dose administered in the current study and for whom pIMDs data were available for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 47
Participants
  Any pIMD(s) | 1
  Related pIMD(s) | 0

23. Secondary Outcome: Number of Participants With Confirmed HZ Cases, as Assessed in the Revaccination Active and Follow-up Phases of the Current ZOSTER-073 Study
Description: as for outcome 6
Time Frame: From Month 24 (pre-revaccination) until Month 49 (24 months post-revaccination Dose 2) in the current ZOSTER-073 study
Population: Analysis was performed on the Exposed Set for revaccination phase, which included all participants with at least one HZ/su revaccination dose administered in the current study and for whom HZ cases data were available for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 47
Participants | 0

24. Secondary Outcome: Number of Participants With Allograft Dysfunction Following Revaccination, as Assessed in the Revaccination Active and Follow-up Phases of the Current ZOSTER-073 Study
Description: Declining allograft function was assessed through all clinically obtained serum creatinine values from 3 months before the first revaccination dose until 3 months after the last revaccination dose. Allograft dysfunction is defined as having a fold increase in serum creatinine of 1.2 greater from the reference timepoint (3 months prior to revaccination).
Time Frame: From Month 24 (pre-revaccination) until Month 37 (12 months post-revaccination Dose 2) in the current ZOSTER-073 study
Population: Analysis was performed on the Exposed Set for revaccination phase, which included all participants with at least one HZ/su revaccination dose administered in the current study and for whom allograft dysfunction following revaccination data were available for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 33
Participants | 4

25. Secondary Outcome: Number of Participants With Allograft Dysfunction Related to Allograft Rejection, as Assessed in the Revaccination Active and Follow-up Phases of the Current ZOSTER-073 Study
Description: Declining allograft function was assessed through all clinically obtained serum creatinine values from 2 months prior to an episode of biopsy-proven rejection and up to 2 months after rejection resolution and cessation of therapeutic immunosuppressive therapy. Allograft dysfunction is defined as having a fold increase in serum creatinine of 1.2 greater from the reference timepoint (2 months prior to an episode of biopsy-proven rejection).
Time Frame: From Month 24 (pre-revaccination) until Month 49 (24 months post-revaccination Dose 2) in the current ZOSTER-073 study
Population: Analysis was performed on the Exposed Set for revaccination phase, which included all participants with at least one HZ/su revaccination dose administered in the current study and for whom allograft dysfunction related to allograft rejection data were available for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 47
Participants | 0

26. Secondary Outcome: Number of Participants With Allograft Dysfunction Related to HZ Episodes, as Assessed in the Revaccination Active and Follow-up Phases of the Current ZOSTER-073 Study
Description: Declining allograft function was assessed through all clinically obtained serum creatinine values from 2 months prior to an episode of HZ and up to 2 months after HZ resolution. Allograft dysfunction is defined as having a fold increase in serum creatinine of 1.2 greater from the reference timepoint (2 months prior to an episode of HZ).
Time Frame: From Month 24 (pre-revaccination) until Month 49 (24 months post-revaccination Dose 2) in the current ZOSTER-073 study
Population: Analysis was performed on the Exposed Set for revaccination phase, which included all participants with at least one HZ/su revaccination dose administered in the current study and for whom allograft dysfunction related to HZ episodes data were available for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group
Number analyzed (Participants) | 47
Participants | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs: Within 7 days after any revaccination; Unsolicited AEs: Within 30 days after any revaccination; SAEs and pIMDs: from Month 24 until Month 37; All-cause mortality, Related SAEs and biopsy-proven allograft rejections: from Day 1 until Month 49, in the current ZOSTER-073 study.
Description: As pre-specified in Protocol, events presented in the All-cause mortality and Serious Adverse Events modules were assessed in both non-revaccinated and revaccinated participants from the Enrolled Set during the specified time frames.
  In the current ZOSTER-073 study, only revaccinated participants from the Exposed Set had their events in the Other Adverse Events module assessed during the specified time frames, and non-serious adverse events were not assessed in non-revaccinated participants.
Arm/Group | HZ/su Group
All-Cause Mortality (participants affected / at risk) | 7/68
Serious Adverse Events (participants affected / at risk) | 23/68
Other Adverse Events (participants affected / at risk) | 43/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HZ/su Group (N=68)
COVID-19 (Infections and infestations) | 6 (8)
Klebsiella urinary tract infection (Infections and infestations) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 3 (3)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
COVID-19 Pneumonia (Infections and infestations) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (2)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HZ/su Group (N=47)
Administration site pain (General disorders) | 40 (68)
Fatigue (General disorders) | 31 (50)
Chills (General disorders) | 19 (25)
Administration site swelling (General disorders) | 16 (25)
Administration site erythema (General disorders) | 14 (22)
Pyrexia (General disorders) | 6 (9)
Injection site pruritus (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 26 (41)
Headache (Nervous system disorders) | 27 (39)
Gastrointestinal disorder (Gastrointestinal disorders) | 16 (21)
Constipation (Gastrointestinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3)
Onychomycosis (Infections and infestations) | 1 (1)
Blindness (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT04176939/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT04176939/SAP_003.pdf